CLINICAL TRIAL: NCT00688636
Title: Infliximab for the Prevention of Recurrent Crohn's Disease After Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Principal Investigator, Miguel Regueiro, Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: C0168X75
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: infliximab
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: infliximab — 5 mg/kg IV at baseline, 2 weeks, 6 weeks and then every 8 weeks x 6
  Other Names: Remicade
  Arms: 1
Drug: placebo — placebo IV at baseline, 2 weeks, 6 weeks and then every 8 weeks x 6
  Arms: 2

SUMMARY:
A randomized, placebo-controlled pilot study to determine endoscopic recurrence of Crohn's disease 12 months after curative, resective ileal or ileocolonic surgery in patients receiving post-operative infliximab or placebo

ELIGIBILITY:
Inclusion Criteria:

* men/women > 18 years of age
* curative resection/ileocolonic anastomosis for Crohn's disease
* may have received previously received infliximab
* if on oral aminosalicylates or corticosteroids, dose must be stable for 4 weeks prior to surgery
* if on 6-mercaptopurine,azathioprine or methotrexate,individual must have been on it for minimum of 3 months prior to surgery with stable dose for 4 weeks
* men and women must use adequate birth control for duration of study and for 6 months after receiving the last infusion
* antibiotics for treatment of Crohn's disease must be discontinued within 12 weeks after surgery; antibiotics are allowable throughout study as long as primary purpose of antibiotic therapy is not for primary treatment of Crohn's disease
* screening lab results must meet screening criteria (hemoglobin = or > 8.5g/dL; Serum glutamic oxaloacetic transaminase ,3 times upper normal limit,platelets =or> 100 x 10 9th/L; lymphocytes count =or> 0.5 x 10 9th/L and neutrophils =or> 1.0 x 10 9th/L
* have a documented negative reaction to a purified protein derivative skin test performed within 3 months prior to baseline
* have a normal chest radiograph results within 3 months prior to baseline
* are capable of providing written informed consent and obtained prior to conducting any protocol-specified procedures
* willing to adhere to the study visit schedule and other protocol requirements
* are considered eligible according to the tuberculosis eligibility assessment, screening and early detection of reactivation rules
* patients who undergo resective surgery and primary ileocolonic anastomosis with a temporary ileostomy upon takedown of the diverting ileostomy.

Exclusion Criteria:

* patients with greater than 10 years of Crohn's disease requiring first resection of a short (<10cm) fibrostenotic stricture
* macroscopically active disease at anastomosis at time of surgery
* presence of stoma
* prior severe infusion reaction to infliximab
* history of anaphylaxis to murine products or other chimeric proteins
* any of the following medications taken within 12 weeks of surgery: cyclosporine, tacrolimus, sirolimus, mycophenolate mofetil, investigational drugs, or medications targeted at reducing tumor necrosis factor
* have a positive stool culture for enteric pathogens, pathogenic ova or parasites, or Clostridium difficile toxin and have clinically significant signs of an enteric infection at screening
* women who are pregnant, nursing or planning pregnancy during the trial or within 6 months after the last infusion
* patient with active tuberculosis, patient newly diagnosed with latent tuberculosis who's receiving tuberculosis prophylaxis, patient with recent close contact to individual with active tuberculosis
* have or have had opportunistic infection within 6 months of screening
* have chest radiograph within 3 months prior to screening that shows malignancy, infection, or abnormalities suggestive of tuberculosis
* documentation of seropositive for HIV
* documentation of a positive test for hepatitis B surface antigen or a history of documented hepatitis C
* have current signs/symptoms of systemic lupus erythematosus, or severe progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic or cerebral diseases
* presence of a transplanted solid organ (with exception of corneal transplant > 3 months prior to randomization)
* Have any current or known malignancy or have history of malignancy within 5 years of screening(except for squamous or basal cell carcinoma of the skin that has been fully excised with no evidence of recurrence)
* have history of lymphoproliferative disease or splenomegaly
* have known substance abuse(drug/alcohol)/dependency within the previous 3 years, history of noncompliance with medical regimens, or other condition that may interfere with adherence to protocol requirements
* are unwilling/unable to undergo multiple venipunctures because of poor tolerability or lack of easy access
* known history of demyelinating disease
* a chronic or recurrent infectious disease
* serious infection, hospitalization for infection, or treatment with IV antibiotics for infection within 2 months prior to randomization
* a serious concomitant illness that may interfere with participation in trial
* concomitant diagnosis/history of congestive heart failure
* current use of prescription doses or chronic/frequent use of non-steroidal anti-inflammatory drugs
* ulcerative colitis
* concurrent participation in another investigative trial
* use of any investigational drug within 30 days prior to randomization

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel D Regueiro, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Regueiro M, Schraut W, Baidoo L, Kip KE, Sepulveda AR, Pesci M, Harrison J, Plevy SE. Infliximab prevents Crohn's disease recurrence after ileal resection. Gastroenterology. 2009 Feb;136(2):441-50.e1; quiz 716. doi: 10.1053/j.gastro.2008.10.051. Epub 2008 Oct 31. PMID 19109962

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 2005 and 2007 there were 24 adult patients with ileal or ileocolonic Crohn's disease undergoing resection who participated in the study.
Groups:
- Infliximab: infliximab: 5 mg/kg IV at baseline, 2 weeks, 6 weeks and then every 8 weeks for 54 weeks
- Placebo: placebo: placebo IV at baseline, 2 weeks, 6 weeks and then every 8 weeks for 54 weeks
Period: Overall Study
Arm/Group | Infliximab | Placebo
Started | 11 | 13
Completed | 9 | 12
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infliximab | Placebo | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43.0 [28 to 49] | 32.0 [26 to 45] | 38.0 [27.0 to 47.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Endoscopic Recurrence: the Proportion of Patients in Endoscopic Recurrence at One Year
Description: Endoscopic recurrence was defined as i2,i3,i4. We used the Rutgeerts' Endoscopic Scoring System. Scores as follows i0, no lesions; i1, 5 or fewer aphthous lesions; i2, more than 5 aphthous lesions with normal mucosa between the lesions or skip areas of larger lesions or lesions confined to the ileocolonic anastomosis; i3, diffuse, aphthous ileitis with diffusely inflamed mucosa; and i4, diffuse inflammation with large ulcers, nodules, and/or narrowing. Endoscopic recurrence was defined as i2,i3,i4 and endoscopic remission was defined as i0 or i1.
Time Frame: one year
Population: The proportion of patients with endoscopic recurrence (> or = i2) at 1 year after surgery
Measure: Number; unit: participants
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 13
participants | 1 | 11
Statistical Analysis 1: Comparison: Infliximab vs Placebo; Test type: Superiority or Other; p = .0005, Fisher Exact

2. Secondary Outcome: Clinical Recurrence at One Year: Defined by Crohn's Disease Activity Index (CDAI) > 200
Description: The Crohn's Disease Activity Index (CDAI) is calculated by a measurement of symptoms, signs, and lab tests over a time period of the previous 7 days. The CDAI includes: Number of very soft stools; sum of abdominal pain ratings: (0=none, 1= mild, 2=moderate, 3=severe); general well being (0=well, 1=slightly below par, 2=poor, 3=very poor, 4=terrible); Symptoms or findings presumed related to Crohn's disease (present): arthritis or arthralgia, iritis or uveitis, erythema nodosum, pyoderma gangrenosum, aphthous stomatitis, anal fissure, fistula or perirectal abscess, other bowel related fistula, febrile episode over 100 degrees during past week, taking lomotil or opiates for diarrhea, abnormal mass (0=none; 0.4=questionable; 1=present) hematocrit [(typical-current) X 6] Normal average male = 47, female =42, body weight
Time Frame: One year
Population: CDAI score > 200
Measure: Number; unit: participants
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 13
participants | 0 | 5

3. Secondary Outcome: Histological Recurrence of Crohn's Disease as Determined From Biopsies of Neo-terminal Ileum Above the Ileocolonic Anastomosis
Description: Histologic recurrence based on a histologic activity score and the presence of polymononuclear cells. The maximum score is 14 per biopsy site.
Time Frame: One year
Population: Histologic activity score
Measure: Number; unit: participants
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 13
participants | 3 | 11

4. Secondary Outcome: C-reactive Protein Concentration as a Surrogate Marker of Inflammation
Description: The CRP was obtained at each study visit as a surrogate marker of inflammation. The CRP was recorded as milligram per deciliter (mg/dl). A normal CRP was 0-0.8 mg/dl; levels exceeding 0.8 mg/dl indicated inflammation.
Time Frame: one year
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 13
mg/dL | 0.5 [0.05 to 0.8] | 0.6 [0.2 to 1.5]

5. Secondary Outcome: Mean Erythrocyte Sedimentation Rate
Description: erythrocyte sedimentation rate value - blood test
Time Frame: one year
Measure: Median (Full Range); unit: mm/h
Arm/Group | Infliximab | Placebo
Number analyzed (Participants) | 11 | 13
mm/h | 30 [10 to 40] | 19 [9 to 34]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Infliximab | Placebo
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/13
Other Adverse Events (participants affected / at risk) | 7/11 | 11/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=11) | Placebo (N=13)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=11) | Placebo (N=13)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Lung nodules (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
partial small-bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
pyleonephritis (Infections and infestations) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 1 (1)
lupus-like reaction (Immune system disorders) | 1 (1) | 0 (0)
abcess (Infections and infestations) | 1 (1) | 1 (1)
crohn's disease exacerbation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infusion reaction (Immune system disorders) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations to our study included a small sample size, a disproportionate number of smokers in the infliximab group, more patients on immunomodulators in the placebo group, and inclusion of patients who had previously received infliximab.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No